CLINICAL TRIAL: NCT06311435
Title: Utilizing Novel Blood RNA Biomarkers as a Diagnostic Tool in the Identification of Long COVID-19
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MaxWell Clinic, PLC (Industry)
Responsible Party: Principal Investigator, Cale T Queen, Executive Director, MaxWell Clinic, PLC
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: FBB-RNA-004
Record Dates: First submitted 2024-03-12; First posted 2024-03-15 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Long COVID
Keywords: COVID-19; Long COVID; Long Haul COVID; Long COVID-19; Long Haul COVID-19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: Participants will be placed into one of fourteen possible cohorts based on their presenting complaints.
Who Masked: Participant
Masking Description: Patients will be assigned a random number from the electronic health record. The only information shared with the sponsor will be Pt ID number, age, gender and state of residence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Participants never infected by SARS-COV-2 (Active Comparator): Participants with no history of SARS-COV-2 infection. This is a control arm of the study. Participants will complete an ethnic survey, medical history survey and undergo two blood draws.
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants with SARS-COV-2 post-infection without long COVID (Active Comparator): Participants with a history of SARS-COV-2 infection, but never developed long term sequalae. This is a control arm of the study. Participants will complete an ethnic survey, medical history survey and undergo two blood draws.
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants with long COVID and current/active respiratory symptoms (Active Comparator): Participants with a history of SARS-COV-2 infection and developed long term sequalae associated with their respiratory system: continued shortness of breath, etc.. This is an experimental arm of the study. Participants will complete an ethnic survey, medical history survey and undergo two blood draws.
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants with long COVID and current/active neurological symptoms (Active Comparator): Participants with a history of SARS-COV-2 infection and developed long term sequalae associated with their neurologic system: brain fog, confusion, etc.. This is an experimental arm of the study. Participants will complete an ethnic survey, medical history survey and undergo two blood draws.
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants who have long COVID with current/active both respiratory and neurological symptoms (Active Comparator): Participants with a history of SARS-COV-2 infection and developed long term sequalae associated with both their respiratory system and their neurologic system. This is an experimental arm of the study. Participants will complete an ethnic survey, medical history survey and undergo two blood draws.
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants who have other current/active long COVID symptoms (Active Comparator): Participants with a history of SARS-COV-2 infection and developed long term sequalae not associated with respiratory or neurological conditions.
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants with neurological symptoms prior to 1 November 2019 without SARS-COV-2 infection (Active Comparator): Participants without a history of SARS-COV-2 infection and had neurological conditions prior to 1 November 2019.
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants with respiratory symptoms before 1 November 2019 w/o SARS-COV-2 prior to 1 Nov 2019 (Active Comparator): Participants without a history of SARS-COV-2 infection and had respiratory conditions prior to 1 November 2019.
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants with neurological symptoms prior to 1 November 2019 with SARS-COV-2 infection (Active Comparator): Participants with a history of SARS-COV-2 infection and had neurological conditions prior to 1 November 2019.
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants with respiratory symptoms prior to 1 November 2019 with SARS-COV-2 infection (Active Comparator): Participants with respiratory symptoms prior to 1 November 2019 with SARS-COV-2 infection
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants with resolved long COVID respiratory symptoms (Active Comparator): Participants with a history of SARS-COV-2 infection and long term respiratory symptoms that have resolved
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants with resolved long COVID neurological symptoms (Active Comparator): Participants with a history of SARS-COV-2 infection and resolved long COVID neurological symptoms
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants with resolved long COVID respiratory and neurological symptoms (Active Comparator): Participants with history of SARS-COV-2 and resolved long COVID respiratory and neurological symptoms
  Interventions: Diagnostic Test: RNA Biomarker Blood Test
- Participants with other resolved long COVID symptoms (Active Comparator): Participants with a history of SARS-COV-2 and other resolved long COVID symptoms
  Interventions: Diagnostic Test: RNA Biomarker Blood Test

INTERVENTIONS:
Diagnostic Test: RNA Biomarker Blood Test — Blood will be collected into a PaxGene Blood tube for processing by sponsor

SUMMARY:
The Primary objective of this study is to determine, using unblinded samples, if it is possible to develop an algorithm for the classification of specific blood RNA from patients with long COVID together and separately from the apparent health normal controls and other medical conditions that share the signs and symptoms of long COVID.

DETAILED DESCRIPTION:
Participants will be screened and provide two blood samples28 (+/- 2) days apart. Based on the participants survey results they will be placed into one of fourteen groups that reflect the type of Long COVID the patient is experiencing. Samples will be shipped to the sponsor who will develop an AI process to validate the type of Long COVID and assess its severity. The long term goal is to develop a reliable test to identify the presence of Long COVID and its severity.

ELIGIBILITY:
Inclusion Criteria:

* Mentally capable of understanding and completing informed consent for the study.
* Precipitants with a lab verified diagnosis of SARS-CoV-2 or clinician note/record that an appropriate rapid test for SARS-CoV-2 was positive.
* To qualify for long COVID group participants will need to have new, persistent symptoms related to SARS-CoV-2 infection. iv. No one under the age of 18.

Exclusion Criteria:

* Subject is unable to provide informed consent.
* Primary Investigator or Sub-Investigator determines the participant's ongoing medical complaints that began after 1 November 2019 are not related to SARS-COV-2 but another disease process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 224 (Estimated)
Dates: Start 2024-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Develop algorithm to classify RNA sequences to identify long COVID | 30 days
  The Primary objective of this study is to determine, using unblinded samples, if it is possible to develop an algorithm for the classification of specific blood RNA from patients with long COVID together and separately from the apparent health normal controls and other medical conditions that share the signs and symptoms of long COVID

SECONDARY OUTCOMES:
Develop algorithm to subclassify specific RNA sequences to subclassify types of Long COVID | 30 Days
  The secondary objective of this study is to determine if it is possible to develop an algorithm that can subclassify specific blood RNA biomarkers in long COVID patients into various symptom-related subcategories to provide clinically relevant treatment options.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Iowa, Iowa City, Iowa
  - The MaxWell Clinic, Brentwood, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided
The results will be published if the hypothesis is supported.